CLINICAL TRIAL: NCT05080686
Title: The Management and Assessment of Pain Control in Rib Fracture With Non-invasive Stabilization: a Randomized Controlled Trial
Brief Title: The Pain Control in Rib Fracture With Non-invasive Stabilization (RCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110-079-F
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-10

CONDITIONS: Rib Fractures; Pain; Thorax; Fracture
Keywords: Rib fractures; pain control; Posthorax Thoraxbelt
MeSH Terms: conditions — Rib Fractures; Pain; Fractures, Bone; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The surgeon will not know the patients' group before or during the surgery. The outcome assessor will not know the group during the whole research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ThoraxBelt (Inpatients) (Experimental): Received ThoraxBelt after the surgery in addition to oral analgesics. Standard care for pain management will be the same as the Standard Care Arm (Inpatients).
  Interventions: Device: Posthorax Thoraxbelt
- Standard Care (Inpatients) (No Intervention): Standard Care with IV PCA and on-request oral painkiller.
- ThoraxBelt (Outpatients) (Experimental): Received ThoraxBelt at the emergency room in addition to oral analgesics. Standard care for pain management will be the same as the Standard Care Arm (Outpatients).
  Interventions: Device: Posthorax Thoraxbelt
- Standard Care (Outpatients) (No Intervention): Standard Care and on-request oral painkiller.

INTERVENTIONS:
Device: Posthorax Thoraxbelt — The patients will be assisted to put on the ThoraxBelt after surgery or at the emergency room by our research members and will be asked to keep it on except for showering through the whole study period.
  Arms: ThoraxBelt (Inpatients); ThoraxBelt (Outpatients)

SUMMARY:
Brief summary:

Background: Rib fractures are one of the most common causes of trauma disabilities and have become an important health issue. Patients usually suffer from severe pain. A rapid and adequate pain control is considered as a priority to improve respiratory mechanics and reduce the risk of pulmonary and systemic complications. So far, there was no gold standard regarding pain control for rib fractures.

Objective: To assess the effect of the newly-designed Prosthorax Thoraxbelt in addition to oral analgesics on pain control of rib fractures

Method: There will be two groups of patients in this study. One group will be the patients with rib fractures who are necessary for in-hospital intense pain control. The other will consist of follow-up patients with rib fractures at an outpatient clinic. The investigators will aim to recruit 30 and 82 patients respectively.

DETAILED DESCRIPTION:
The study has been approved by the hospital research ethics committee.

Arm1: The management and assessment of pain control in rib fracture with non-invasive stabilization: a randomized controlled trial (inpatients)

Arm2: The management and assessment of pain control in rib fracture with non-invasive stabilization: a randomized controlled trial (outpatients)

Primary outcome:

1. inpatient: Visual analog scale (VAS) for 6 hours, 12 hours and 24 hours after the surgery
2. outpatient: Visual analog scale (VAS) for the times at emergency room; 3 days, 3 weeks and 3 months after rib fracture at an outpatient clinic.

Secondary outcome:

* inpatients

  1. The accumulated dose of the inter-venous patient-controlled analgesic drug within 6 hours, 24 hours and 48 hours after the surgery
  2. Complication during the hospital stay
  3. Hospital stay
  4. VAS before discharge
  5. Unanticipated events (ICU admission, a second surgery, death)
  6. VAS during the 1-week, 1-month and 3-month outpatient clinic visit after the surgery
  7. An X-ray examination at an outpatient clinic
  8. Compliance on ThoraxBelt after discharge
* outpatients

  1. Complication during the follow-up period
  2. Unanticipated events (ward admission, ICU admission, a surgery, OHCA)
  3. Compliance on ThoraxBelt after discharge
  4. An X-ray examination at an outpatient clinic

ELIGIBILITY:
Inclusion Criteria:

* The adult patients with rib fractures (inpatients/outpatients)
* The patients will be assessed to the further admission (inpatients)
* The patients will be assessed to be at follow-up clinic visit (outpatients)

Exclusion Criteria:

* The accident of rib fractures has been occurred over 24 hours. (inpatients/outpatients)
* Refuse to be arranged to the admission (inpatients)
* Refuse to receive the CT scan (inpatients/outpatients)
* Chest wall infection or other diseases (inpatients/outpatients)
* Chest wall infected by rumors (inpatients/outpatients)
* Pregnancy (inpatients/outpatients)
* Further complications arise (inpatients/outpatients)
* Known allergy to ThoraxBelt (inpatients/outpatients)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Inpatients: Visual analog scale (VAS) | 48 hours
  A pain score will be assessed to each patient after the total amount of visual analog scale. The minimum is 0 and the maximum is 10, from the least pain to the highest pain.
Outpatients: Visual analog scale (VAS) | 3 months
  A pain score will be assessed to each patient after the total amount of visual analog scale. The minimum is 0 and the maximum is 10, from the l

SECONDARY OUTCOMES:
Inpatients: IV PCA dose | 48 hours
  the accumulated IV PCA drug dose
Inpatients: On-request oral painkiller dose | 48 hours
  the accumulated oral painkiller dose
Inpatients: Complication during the hospital stay | 48 hours
  Any complications whether related to ThoraxBelt or not
Inpatients: Length of hospital stay | 1 month
  the amount of days in hospital stay
Inpatients: VAS before discharge | 3 months
  Visual analog scale before discharge
Inpatients: The amount of unanticipated events | 3 months
  send to the ICU admission, a second surgery or death
Inpatients: VAS in outpatient clinic follow-up | 3 months
  VAS during the 1-week, 1-month and 3-month outpatient clinic visit after the surgery
Inpatients/Outpatients: X-ray examination | 3 months
  An X-ray examination at an outpatient clinic
Inpatients/Outpatients: Compliance on ThoraxBelt after discharge | 3 months
  How long is the ThroaxBelt removed except during the bath within the whole day. The unit is hour.
Outpatients: Complication during the follow-up period | 6 months
  Any complications whether related to ThoraxBelt or not
Outpatients: The amount of unanticipated events | 3 months
  send to the ward admission, ICU admission, a surgery or OHCA

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently, we have no plan on sharing the IPD.